CLINICAL TRIAL: NCT04756609
Title: Evaluation of the Benefit of a Systematic Offer of Nurse-Driven SARS-Cov2 Screening by Rapid Testing in Emergency Departments in the Paris Metropolitan Area
Brief Title: Systematic Offer of Nurse-Driven Screening for COVID-19 in Emergency Departments in the Paris Metropolitan Area, DEPIST-COVID
Acronym: DEPIST-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: APHP201625; IDRCB: 2020-A03532-37 (Other: ANSM)
Record Dates: First submitted 2021-02-06; First posted 2021-02-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: SARS-CoV Infection; Nurse's Role
Keywords: SARS-CoV-2; Mass screening; Emergency service; hospital Nurses; Prevention and control
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic offer of nurse-driven SARS-CoV-2 screening + usual practice (Experimental): Systematic offer of nurse-driven SARS-CoV-2 screening combined with usual practice
  Interventions: Procedure: Systematic offer of nurse-driven SARS-CoV-2 screening combined with usual practice
- Control group: Usual emergency department practice (Active Comparator): Usual emergency department practice with physician-directed diagnostic testing
  Interventions: Other: Usual emergency department practice with physician-directed diagnostic testing

INTERVENTIONS:
Procedure: Systematic offer of nurse-driven SARS-CoV-2 screening combined with usual practice — I- A SARS-CoV2 self-administered questionnaire about SARS-CoV2 symptoms, possibilities of close contacts, risk exposure situations and socio-demographic characteristics will be offered to patients included who are capable of filling it out.
  * The patient will fill out the questionnaire and hand it in to the nurse caring for him/her.
  * The nurse, regardless of the answers to the questionnaire, will offer the SARS-CoV2 screening.
  * A nasopharyngeal swab for SARS-CoV2 will be carried out.
  * A patient will be considered as symptomatic if he/she presents one or more symptoms listed in the questionnaire.
  * For symptomatic patients, a SARS-CoV2 for multiplex PCR will be carried out. This analysis takes 75 minutes.
  * For asymptomatic patients, a RT-LAMP test will be carried out. This analysis takes 5 to 15 minutes.
  Arms: Systematic offer of nurse-driven SARS-CoV-2 screening + usual practice
Other: Usual emergency department practice with physician-directed diagnostic testing — The physician offers a SARS-CoV2 test according to current recommendations. The tests are prescribed as a means of diagnosis for patients presenting symptoms suggestive of Covid-19 or as a means of diagnosis for patients requiring hospitalisation for another cause, before their transfer to hospital. Patients will be cared for according to usual procedures of each hospital. Patients tested positive will be asked to fill out the DEPIST-COVID questionnaire. Patients who had not completed it will be contacted by phone to answer the questions over the phone.
  Arms: Control group: Usual emergency department practice

SUMMARY:
European countries faced another wave of the SARS-CoV2 pandemic, which has led to a second lockdown in France in November 2020 in order to avoid overwhelming health services. To prevent or reduce another wave, the strategy calls for vaccination, maintaining barrier measures and testing and isolating infected persons in order to break the cycles of infection. The latter objective is made difficult by the existence of asymptomatic carriers or symptomatic carriers that have very few symptoms and that aren't tested. Identification of these carriers in the general population is usually based on a search for close contact persons from those who were tested positive or from identified clusters.

Experiments of mass testing are being carried out or were carried out, for example in Liverpool or Slovakia but, in order for them to be effective, they must be repeated, which limits feasibility. Another strategy of wide screening in the general population to identify asymptomatic persons is to offer a systematic screening during medical consultations and particularly in the emergency departments (ED). This strategy grants access to the entire population attending health facilities, including persons with lower income. This strategy can be conducted continuously in order to: 1) contribute to controlling the epidemic by identifying and isolating asymptomatic persons and their close contacts; 2) provide an observatory on the evolution of viral circulation in the general population.

To the best the knowledge, this strategy has not been evaluated and will be tested it in 18 emergency departments in the Paris Metropolitan area, one of the most SARS-CoV2 affected regions.

The aim is to evaluate the benefit of a systematic offer of SARS-Cov2 screening by rapid testing (molecular multiplex PCR/ RT-LAMP) to identify infected persons, associated with the usual practice of the EDs (intervention strategy) compared to a period based on usual practice of the EDs (control strategy)

The strategies will be compared during two periods following a cluster-randomized two-period crossover design.

During intervention periods, nurses will suggest performing a SARS-CoV2 test to patients using a PCR multiplex for symptomatic patients and a RT-LAMP for asymptomatic patients.

DETAILED DESCRIPTION:
European countries faced another wave of the SARS-CoV2 pandemic, which has led to a lockdown in France in November 2020 in order to avoid overwhelming health services. To prevent or reduce another wave, the strategy calls for vaccination, maintaining barrier measures and testing and isolating infected persons in order to break the cycles of infection. The latter objective is made difficult by the existence of asymptomatic carriers or symptomatic carriers that have very few symptoms and that aren't tested. Identification of these carriers in the general population is usually based on a search for close contact persons from those who were tested positive or from identified clusters.

Experiments of mass testing are being carried out or were carried out, for example in Liverpool or Slovakia but, in order for them to be effective, they must be repeated, which limits feasibility. Another strategy of wide screening in the general population to identify asymptomatic persons is to offer a systematic screening during medical consultations and particularly in the emergency departments (ED). This strategy grants access to the entire population attending health facilities, including persons with lower income. This strategy can be conducted continuously in order to: 1) contribute to controlling the epidemic by identifying and isolating asymptomatic persons and their close contacts; 2) provide an observatory on the evolution of viral circulation in the general population.

To the best of the knowledge, this strategy has not been evaluated and will be tested it in 18 emergency departments in the Paris Metropolitan area (Ile-de-France), one of the most SARS-CoV2 affected regions.

The primary objective is to evaluate the benefit of a systematic offer of nurse-driven SARS-Cov2 screening by rapid testing (molecular multiplex PCR/ RT-LAMP) to identify infected persons, associated with the usual practice of the EDs (intervention strategy) compared to a period based on usual practice of the EDs (control strategy).

The primary outcome is the proportion of patients tested positive for SARS-CoV2 amongst the flow of consulting adults.

The secondary outcomes are to:

* compare the proportion of patients tested positive for SARS-CoV2 amongst asymptomatic patients tested in the Paris Metropolitan area at the same period (the comparison will also be done amongst the geographical area of each ED, amongst symptomatic patients tested and also amongst the entire tested population)
* evaluate the feasibility of the screening strategy
* describe the patients tested for SARS-Cov2 in both periods :
* proportion of positive tests
* proportion of asymptomatic patients amongst tested patients and amongst SARS-Cov2 positive patients
* For the symptomatic patients tested positive : symptomology
* Patient exposure factors with the DEPIST-COVID questionnaire and according to SARS-Cov2 test result.
* describe socio-demographic and behavioral factors and habits associated with SARS-Cov2 infection in patients tested in one of the following schemes: DEPIST-COVID, ComCor (Pasteur Institute) and COVISAN.
* estimate the incidence of new SARS-Cov2 infections in the Paris Metropolitan area: proportion of positive patients and their profiles. To estimate the under-detection of cases in the region, and compare with results from the model experiment.
* estimate the number of close contact persons who have been tested for SARS-Cov2, who have been tested positive and who have been isolated over both periods.

Methods The strategies will be compared during two periods in 18 EDS of Paris metropolitan area following a cluster-randomized two-period crossover design. Each period will last 1 month. Patients will participate to a follow-up call (within 15 days ±10). The periods will be separated by an expected period of washout of a minimum of 1 day .

During intervention periods, nurses will suggest performing a SARS-CoV2 test to patients. According to the answers to a self-administered questionnaire, a PCR multiplex will be performed for symptomatic patients and a RT-LAMP for asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

All consulting adults visiting a participating ED

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138352 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients tested positive for SARS-CoV2 amongst the flow of consulting adults | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)

SECONDARY OUTCOMES:
Proportion of positive patients amongst asymptomatic patients and in the Paris Metropolitan area at the same period (these proportions will be compared amongst each ED geographic area, amongst symptomatic patients and amongst the tested population) | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)
Feasibility of screening strategy : proportion of patients having completed the questionnaire, proportion of tests offered , accepted and performed, proportion of patients notified of the result and staff involved | At the end of the expected duration of the study (2 months and 15±10 days + wash out in each ED)
Description of patients tested in both periods (proportion of positive tests and of asymptomatic patients) | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)
For symptomatic patients: description of the symptomatology | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)
Description of patients tested in both periods: patient exposure factors with the DEPIST-COVID questionnaire | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)
Sociodemographic, behavioural factors and habits associated with SARS-Cov2 infection in patients tested in the following schemes: DEPIST-COVID, ComCor and COVISAN . | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)
Incidence of SARS-Cov2 infections in Paris Metropolitan area : proportion of positive patients and their profiles. To estimate the under-detection of cases in the region, and compare with results from the model experiment . | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)
Number of close contact persons who have been tested for SARS-Cov2, who have been tested positive and who have been isolated over both periods. | At the end of the expected duration of the inclusion period (an average of 3 months in each ED)

CONTACTS AND LOCATIONS:
Overall Officials: Judith LEBLANC, RN, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- URC-EST, Hôpital saint-Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No
The study data are owned by the Assistance Publique - Hôpitaux de Paris (AP-HP) sponsor, "Département de la Recherche Clinique et du Développement". The data are not freely available.
  No data may be transmitted unless a contract has first been signed between the AP-HP and an external partner interested in the data.
  For all inquiries, please contact the following:
  DJENNAOUI Fatiha <fatiha.djennaoui@aphp.fr> and [DRC] Secretariat Promotion Délégation à la Recherche Clinique et à l'Innovation <drc-secretariat-promotion@aphp.fr>.

REFERENCES:
- [Derived] Leblanc J, Dusserre-Telmon L, Chauvin A, Simon T, Sabbatini CE, Hemming K, Colizza V, Berard L, Convert J, Lazazga S, Jegou C, Taibi N, Dautheville S, Zaghia D, Gerlier C, Domergue M, Larrouturou F, Bonnet F, Fontanet A, Salhi S, LeGoff J, Cremieux AC; DEPIST-COVID group; FHU IMPEC (Improving Emergency Care) group. Intensified screening for SARS-CoV-2 in 18 emergency departments in the Paris metropolitan area, France (DEPIST-COVID): A cluster-randomized, two-period, crossover trial. PLoS Med. 2023 Dec 7;20(12):e1004317. doi: 10.1371/journal.pmed.1004317. eCollection 2023 Dec. PMID 38060611